CLINICAL TRIAL: NCT00302367
Title: An Open Label Phase I/II Study of Dopamine Transporter Receptor Occupancy With OROS and Immediate Release Methylphenidate as Measured With C-11 Altropane in Human Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc. (Industry)
Responsible Party: Thomas J. Spencer, MD, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 2003-p-002058
Record Dates: First submitted 2006-03-10; First posted 2006-03-14 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2011-07

CONDITIONS: Healthy Volunteers

INTERVENTIONS:
Drug: OROS methylphenidate hydrochloride
Drug: immediate release methylphenidate hydrochloride

SUMMARY:
The specific aim of this study is to document the pharmacokinetics of DAT receptor occupancy of OROS and immediate release (IR) MPH using PET scanning with C-11 altropane as the ligand. We hypothesize that the time to maximal receptor occupancy and the degree of receptor occupancy of immediate release (IR) MPH will be shorter and greater (respectively) than with an equipotent dose of OROS MPH.

DETAILED DESCRIPTION:
This protocol seeks to document the pharmacokinetics of DAT receptor occupancy of OROS and immediate release (IR) MPH using PET and C-11 altropane. The main target of MPH in the brain is the dopamine transporter (DAT). We have an exquisitely sensitive methodology to measure DAT occupancy using C-11 Altropane and Positron Emission Tomography (PET). This research will provide novel and unique information toward a better understanding of the mechanism of action of long-acting stimulant formulations to enable new drug development and an estimation of the relative abuse potential of the current formulation.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent to participate in the study.
2. Age: 18 - 55
3. If female, non-pregnant, non-nursing with a negative serum pregnancy test and using an adequate form of birth control.
4. Supine and standing blood pressure within the range 110/60 to 150/90 mmHg.
5. Heart rate, after resting for 5 minutes, within the range 46-90 beats/min.
6. Subjects who are within 20% of the ideal weight for height as
7. Right handed.

Exclusion Criteria:

1. Diagnosis of any psychotic disorder, bipolar disorder, severe depression, severe anxiety, or Autism. Subjects with mild mood, oppositional, conduct, and anxiety disorders may be permitted to participate if considered appropriate by the investigator.
2. Scores of Baseline Scales:

   Hamilton Depression Scale > 17 (out of a possible 67 on the 21-item scale)[18] Beck Depression Inventory > 19 (out of a possible 63 on the 21-item scale)[19] Hamilton Anxiety Scale > 21 (out of a possible 56 on the 14-item scale) [20]
3. Tics or Tourette's Syndrome.
4. History of head trauma with loss of consciousness, organic brain disorders, seizures, or neurosurgical intervention.
5. Any clinically significant chronic medical condition, in the judgment of the investigator.
6. Mental impairment as evidenced by an I.Q. <75.
7. Exposure to dopamine receptor antagonists within the previous three (3) months.
8. Exposure to radiopharmaceuticals within four (4) weeks prior to PET scan.
9. Subjects receiving psychotropic medication.
10. Any clinically significant abnormality in the screening laboratory tests, vital signs, or 11-lead ECG, outside of normal limits.

12. Any woman of childbearing potential who is seeking to become pregnant or suspects that she may be pregnant.

13. Subjects with a known recent history (within the past six (6) months) of illicit drug or alcohol dependence

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20
Dates: Start 2004-01; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
The DAT receptor occupancy of OROS MPH and Metadate CD using PET scanning with C-11 Altropane. Objective measures also provided by d and l ritalinic acid and methylphenidate levels at pre-dose through hour 10.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Spencer, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Cambridge, Massachusetts, United States